CLINICAL TRIAL: NCT07317791
Title: Multicenter Prospective Validation of Cough Flow With Tracheostomy Tube and Speaking Valve (CFsv) >100 L/Min as a Criterion Decannulation Threshold in Prolonged Tracheostomy Patients
Brief Title: Cough Flow as a Criterion Decannulation Threshold in Prolonged Tracheostomy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hongying Jiang, MD (Other)
Responsible Party: Sponsor-Investigator, Hongying Jiang, MD, Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-hxkfzx-dzx-002
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Tracheostomy
Keywords: Decannulation; Cough peak flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decannulation Protocol Group (Experimental): all patients included in the study will undergo standardized decannulation assessment.
  Interventions: Other: standardized tracheostomy decannulation protocol

INTERVENTIONS:
Other: standardized tracheostomy decannulation protocol — Step 1: Confirm that the patient is clinically stable. Step 2: Speaking valve (SV) with transtracheal end-expiratory pressure (TTPEE) measurement.
  Step 3: Measure the CFsv. Step 4: Continue wearing the SV for 4 hours. During this period, suctioning is not performed via the tracheostomy tube.
  Step 5: Assess readiness for decannulation. The CFsv is measured again prior to decannulation. If the value exceeds 100 L/min, decannulation is performed.

SUMMARY:
Background: International studies have proposed a cough peak flow (CPF) of ≥160 L/min as a reference threshold for safe decannulation. However, this measurement requires prior removal of the tracheostomy tube, which is often difficult for Chinese patients and their families to accept due to cultural and safety concerns. Additionally, there is a lack of rapid, user-friendly, and widely applicable quantitative tools in clinical practice within ICUs or rehabilitation specialties in China. Moreover, the heterogeneity among domestic patient populations with different underlying conditions (such as neuromuscular diseases, spinal cord injuries, stroke, and respiratory failure) makes it challenging to apply a single foreign-derived indicator. In our center's prospective study from 2019 to 2022(Respiratory Research 2024;25:128), the investigators proposed and preliminarily validated that a cough flow measured with tracheostomy tube and speaking valve (CFSV) >100 L/min could serve as a threshold for safe decannulation. Among 193 patients with long-term tracheostomy tubes, 105 were decannulated based on this threshold, with a success rate of 98.1%. Only two cases required reintubation within 48 hours (1.9%), and the six-month reintubation rate was 2.9%, which is significantly better than previously reported domestic and international data (reintubation rates of 5-15%). For patients with insufficient CFSV, after an average of 26 days of individualized cough enhancement rehabilitation, 91% achieved the threshold and ultimately succeeded in decannulation. This suggests that 100 L/min may be a more physiologically appropriate threshold for Chinese (and even East Asian) populations with indwelling tracheostomy tubes, and that CFSV combined with systematic rehabilitation interventions can significantly improve decannulation rates. However, these conclusions are derived from single-center data with a limited sample size, and the diversity of diseases and regional variations in medical standards may affect generalizability. Therefore, there is an urgent need for multicenter, large-sample prospective studies to validate the effectiveness, accuracy, and feasibility of CFSV >100 L/min as a quantitative standard for safe decannulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Tracheostomy tube in place for ≥14 days
* Weaned from ventilator for more than 48 hours, or in a state of spontaneous breathing
* Patient and family members have provided informed consent

Exclusion Criteria:

* Severe craniofacial deformity preventing CFsv measurement
* Known obstructive upper airway pathology precluding tracheostomy tube removal
* Laryngopharyngeal trauma
* Inability to tolerate cuff deflation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Decannulation Success | 48 hours post-decannulation
  No requirement for tracheostomy tube reinsertion within 48 hours after decannulation

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, MD, Study Chair — Beijing Rehabilitation Hospital of Capital Medical University
Locations (5):
- China (5):
  - Beijing Rehabilitation Hospital, Capital Medical University, Beijing,China, Beijing, Beijing Municipality
  - Hunan Rehabilitation Hospital, Hunan, Hunan
  - Jiangbin Hospital of Guangxi Zhuang Autonomous Region, Guangxi, Jiangbin
  - YanBian University Hospital, Jilin, Yanbian
  - Zhengzhou Central Hospital Affiliated to Zhengzhou University, Henan, Zhengzhou